CLINICAL TRIAL: NCT04448210
Title: Web-based Resource for Children and Adolescents About Clinical Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Principal Investigator, Alison Parker, Research Scientist, Innovation Research & Training
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R44NR019565 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Chronic Illnesses, Multiple
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational website intervention (Experimental): The intervention is an educational website designed to teach youth (12-17 years) about pediatric clinical trials.
  Interventions: Behavioral: DigiKnowIt News: Teen
- Wait-list control (No Intervention): The wait-list control group did not receive the intervention between the pre-test and post-test assessments. After completing the post-test questionnaire, youth in the wait-list control group had the option to receive access to the intervention (DigiKnowIt News).

INTERVENTIONS:
Behavioral: DigiKnowIt News: Teen — Teens will interact with a multimedia educational website that will teach them about pediatric clinical trials including topics such as participant rights and safety, benefits and costs to participating in a study, and different types of procedures used in trials.
  Arms: Educational website intervention

SUMMARY:
The overall aims of this project are to: 1) create a developmentally appropriate interactive educational website for adolescents called DigiKnowIt News: Teen, and 2) examine the feasibility of DigiKnowIt News: Teen in a small randomized control trial with adolescents.

DETAILED DESCRIPTION:
Youth (N=30) will be recruited to participate in the feasibility study. Parent permission and youth assent will be sought. Participants will be randomized into one of two study arms: intervention and wait-list control. All participants will complete a web-based pre-test questionnaire. Youth in the intervention group will then receive access to DigiKnowIt News: Teen for one week. Approximately one week after completing the pre-test questionnaire, all participants will complete a web-based post-test questionnaire (the post-test for youth in the intervention group will also include Consumer Satisfaction Questions). Youth in the wait-list control group will then receive access to DigiKnowIt News: Teen for one week. After one week, they will complete a Consumer Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 12 and 17 years.
* Participants must have access to a computer or tablet with Internet connection.
* Participants must be able to read and write in English fluently.

Exclusion Criteria:

* Participants must NOT have previously participated in a clinical trial.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2020-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Parker, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Website Intervention | Wait-list Control
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Website Intervention | Wait-list Control | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.14 (1.78) | 14.55 (1.64) | 14.33 (1.71)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 8 | 20
  Female | 10 | 10 | 20
  Non-Binary | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 3 | 3
  White | 18 | 12 | 30
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Baseline Knowledge Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will respond to 25 questions that assess their factual knowledge about clinical research (e.g., Who is part of a clinical trial?). Questions are in multiple choice format and some questions have multiple correct answers. The correct responses were summed across the questions. The range of scores was from 0 to 46. Higher scores indicate more knowledge about clinical research.
  units on a scale | 35.74 (4.96) | 36.25 (4.04) | 36.00 (4.47)
Baseline Attitudes Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to 6 questions that assess their positive attitudes about clinical trials (e.g., How do you feel about kids participating in clinical trials?; 1=Not good at all; 2=Not very good; 3=Not sure; 4=Good; 5=Very good). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5.
  Higher scores indicate more positive attitudes toward clinical trials.
  units on a scale | 3.76 (.75) | 3.85 (.65) | 3.80 (.70)
Baseline Beliefs Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to 5 questions that assess their beliefs about positive aspects of pediatric clinical research (e.g., I believe that clinical trials can help kids; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more positive beliefs about clinical research.
  units on a scale | 4.11 (.64) | 4.21 (.51) | 4.16 (.58)
Baseline Self-Efficacy for Gathering Information Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to 9 questions related to their self-efficacy for making decisions related to participation in clinical trials for gathering information about clinical trials (e.g., How sure are you that you can do the following things: Ask my parents questions for more information about clinical trials?; 1 = I cannot do it at all; 5 = I know I can do it.). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more self-efficacy for gathering information about clinical trials.
  units on a scale | 4.23 (.61) | 4.21 (.52) | 4.22 (.56)
Baseline Self-Efficacy to Communicate Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to 10 questions related to their self-efficacy for making decisions related to participation in clinical trials for communicating about clinical trials (e.g., Tell the researcher that I don't want to participate in the clinical trial, even if they really want me to do it; 1 = I cannot do it at all; 5 = I know I can do it.). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more self-efficacy about communicating about clinical trials.
  units on a scale | 4.49 (.61) | 4.56 (.54) | 4.52 (.57)
Baseline Confidence Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to additional items3 questions to measure youths' confidence for participating clinical trials (e.g., I know what rights I have in a clinical trial. I know whom to ask if I need more information about a clinical trial.; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more confidence for participating in clinical trials.
  units on a scale | 3.39 (.67) | 3.35 (.63) | 3.37 (.64)
Baseline Procedural Fears Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to 4 questions related to their perceptions of fear or anxiety about different types of medical procedures, including getting a needle in the arm, injection in the leg, getting a scan, and taking new medicine, on a 5-point Likert scale (1 = Not at all afraid or anxious, 2 = Somewhat afraid or anxious, 3 = Moderately afraid or anxious, 4 = Very afraid or anxious, 5 = Extremely afraid or anxious). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more fears about medical procedures.
  units on a scale | 2.28 (.75) | 2.46 (.80) | 2.37 (.77)
Baseline Likelihood of Participation Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to one question about the likelihood of participating in a clinical trial (i.e., If you were asked to be in a clinical trial, how likely would you be to participate?) using a 5-point Likert scale (1 = Not likely; 5 = Extremely likely). The minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate increased likelihood of participating in a clinical trial.
  units on a scale | 3.57 (.98) | 3.74 (.81) | 3.65 (.89)
Baseline Fear Preventing Participation Scores [Mean (Standard Deviation); unit: units on a scale] — Youth will be asked to respond to one question about the likelihood of their fear preventing them from participating in a clinical trial (i.e., How likely is it that your fearful or anxious feelings could stop you from participating in a clinical trial in the future?) using a 5-point Likert scale (1 = Not likely; 5 = Extremely likely). The minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate increased likelihood of fear preventing them from participating in a clinical trial.
  units on a scale | 2.29 (.78) | 2.35 (1.09) | 2.32 (.93)

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Scores at 1 Week
Description: Youth will respond to 25 questions that assess their factual knowledge about clinical research (e.g., Who is part of a clinical trial?). Questions are in multiple choice format and some questions have multiple correct answers. The correct responses were summed across the questions. The range of scores is from 0 to 46. Higher scores indicate more knowledge about clinical research.
Time Frame: 1 week
Population: In this study, participants were able to skip questions in the questionnaires. Thus, there may not be complete data for all participants for this outcome.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 19 | 20
units on a scale | 35.32 (1.00) | 36.93 (.94)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p < .25, ANOVA

2. Primary Outcome: Attitudes Scores at 1 Week
Description: Youth will be asked to respond to 6 questions that assess their positive attitudes about clinical trials (e.g., How do you feel about kids participating in clinical trials?; 1=Not good at all; 2=Not very good; 3=Not sure; 4=Good; 5=Very good). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more positive attitudes toward clinical trials.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 22 | 20
units on a scale | 3.92 (.09) | 3.87 (.09)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .72, ANOVA

3. Primary Outcome: Beliefs Scores at 1 Week
Description: Youth will be asked to respond to 5 questions that assess their beliefs about positive aspects of pediatric clinical research (e.g., I believe that clinical trials can help kids; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more positive beliefs about clinical research.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 22 | 20
units on a scale | 4.40 (.09) | 4.23 (.09)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .16, ANOVA

4. Primary Outcome: Self-Efficacy to Communicate Scores at 1 Week
Description: Youth will be asked to respond to 10 questions related to their self-efficacy for making decisions related to participation in clinical trials for communicating about clinical trials (e.g., Tell the researcher that I don't want to participate in the clinical trial, even if they really want me to do it; 1 = I cannot do it at all; 5 = I know I can do it.). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more self-efficacy about communicating about clinical trials.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 22 | 20
units on a scale | 4.59 (.10) | 4.48 (.10)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .43, ANOVA

5. Primary Outcome: Self-Efficacy to Gather Information Scores at 1 Week
Description: Youth will be asked to respond to 9 questions related to their self-efficacy for making decisions related to participation in clinical trials for gathering information about clinical trials (e.g., How sure are you that you can do the following things: Ask my parents questions for more information about clinical trials?; 1 = I cannot do it at all; 5 = I know I can do it.). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more self-efficacy for gathering information about clinical trials.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 22 | 20
units on a scale | 4.33 (.09) | 4.38 (.09)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .69, ANOVA

6. Primary Outcome: Confidence Scores at 1 Week
Description: Youth will be asked to respond to 3 questions to measure youths' confidence for participating clinical trials (e.g., I know what rights I have in a clinical trial. I know whom to ask if I need more information about a clinical trial.; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more confidence for participating in clinical trials.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 22 | 20
units on a scale | 3.91 (.14) | 3.73 (.14)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .38, ANOVA

7. Primary Outcome: Procedural Fears Scores at 1 Week
Description: Youth will be asked to respond to 4 questions related to their perceptions of fear or anxiety about different types of medical procedures, including getting a needle in the arm, injection in the leg, getting a scan, and taking new medicine, on a 5-point Likert scale (1 = Not at all afraid or anxious, 2 = Somewhat afraid or anxious, 3 = Moderately afraid or anxious, 4 = Very afraid or anxious, 5 = Extremely afraid or anxious). Responses to this scale were averaged and the minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate more fears about medical procedures.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 22 | 20
units on a scale | 2.25 (.10) | 2.24 (.10)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .94, ANOVA

8. Primary Outcome: Likelihood of Participation Scores at 1 Week
Description: Youth will be asked to respond to one question about the likelihood of participating in a clinical trial (i.e., If you were asked to be in a clinical trial, how likely would you be to participate?) using a 5-point Likert scale (1 = Not likely; 5 = Extremely likely). The minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate increased likelihood of participating in a clinical trial.
Time Frame: 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 21 | 19
units on a scale | 3.63 (.15) | 3.65 (.15)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .94, ANOVA

9. Primary Outcome: Fear Preventing Participation Scores at 1 Week
Description: Youth will be asked to respond to one question about the likelihood of their fear preventing them from participating in a clinical trial (i.e., How likely is it that your fearful or anxious feelings could stop you from participating in a clinical trial in the future?) using a 5-point Likert scale (1 = Not likely; 5 = Extremely likely). The minimum scale score was 1 and the maximum scale score was 5. Higher scores indicate increased likelihood of fear preventing them from participating in a clinical trial.
Time Frame: 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-list Control
Number analyzed (Participants) | 21 | 20
units on a scale | 2.13 (.18) | 2.40 (.18)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-list Control; Test type: Superiority; p = .30, ANOVA

ADVERSE EVENTS:
Time Frame: From baseline to end of intervention at 1 week
Description: The participants in the study completed web-based questionnaires and utilized an educational website (if in the intervention group). The risks associated with this study were minimal and the participants were not at risk for mortality as a function of participating in this study. Because this study investigated an online behavioral intervention, All-Cause Mortality was not monitored or assessed.
Groups:
- Wait-list Control: This is a wait-list control group and they did not receive an intervention.
Arm/Group | Educational Website Intervention | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT04448210/Prot_SAP_000.pdf